CLINICAL TRIAL: NCT01560936
Title: Surveillance Study of Bacterial Contamination of the Parent's Cell Phone in the NICU and the Effectiveness of an Antimicrobial Gel in Reducing Transmission to the Hands
Brief Title: Surveillance Study of Bacterial Contamination of the Parent's Cell Phone in the NICU
Status: Completed | Type: Observational
Sponsor: Pediatrix (Other)
Responsible Party: Sponsor
Other Study IDs: 3.0
Record Dates: First submitted 2012-03-19; First posted 2012-03-22 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2013-05

CONDITIONS: Bacterial Contamination Rate of the Cell Phones
Keywords: bacterial contamination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the contamination rate of the parents cell phone in a newborn intensive care setting and identify the types of bacteria contaminating the cell phone as well as evaluating the effectiveness of an antimicrobial gel in reducing the transmission of bacteria from the cell phone to the parents hands.

DETAILED DESCRIPTION:
J Perinatol. 2013 Dec;33(12):960-3. doi: 10.1038/jp.2013.108. Epub 2013 Sep 5.

ELIGIBILITY:
Inclusion Criteria:

* Parents with a cell phone

Exclusion Criteria:

* Parents that do not have a cell phone

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Parent's that have a cell phone when visiting their child in the NICU.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Determine contamination rate of parents cellphone in the NICU and identify types of bacteria on cell phones while evaluating the effectiveness of antimicrobial gel in reducing the transmission of bacteria from cellphone to parents hands. | contamination rate through bacterial swabs

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kamitsuka, MD, Principal Investigator — Swedish Hospital and Medical Center
Locations (1):
- Swedish Medical Center, Seattle, Washington, United States